CLINICAL TRIAL: NCT04587206
Title: An Open Label, Randomized, Single Dose, 2-sequence, 4-period, Cross-over Clinical Trial to Evaluate the Pharmacokinetics and Tolerability of CKD-348 With Co-administration of CKD-828, D097 and D337 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Evaluate the Pharmacokinetics and Tolerability of CKD-348
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A86_06BE2007
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Hypertension and Dyslipidemia
Keywords: CKD-348
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Sequence 1 (Experimental): Period 1: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Period 2: CKD-348- A single oral dose of 1 tablet under fasting condition
  Period 3: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Period 4: CKD-348- A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-348; Drug: CKD-828, D097, D337
- Experimental: Sequence2 (Experimental): Period 1: CKD-348- A single oral dose of 1 tablet under fasting condition
  Period 2: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Period 3: CKD-348- A single oral dose of 1 tablet under fasting condition
  Period 4: CKD-828, D097, D337- A single oral dose of 3 tablets under fasting condition
  Interventions: Drug: CKD-348; Drug: CKD-828, D097, D337

INTERVENTIONS:
Drug: CKD-348 — QD, PO
Drug: CKD-828, D097, D337 — QD, PO

SUMMARY:
A Clinical Trial to evaluate the Pharmacokinetics and Tolerability of CKD-348

DETAILED DESCRIPTION:
A Phase 1 Clinical Trial to evaluate the tolerability and pharmacokinetics in healthy adult volunteers after administration of CKD-348 and co-administration of CKD-828, D097, D337.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 years
2. Weight ≥50kg (man) or 45kg (woman), with calculated body mass index (BMI) of 18 to 30 kg/m2
3. Those who meet the blood pressure criteria during screening tests:

   A. Systolic Blood Pressure: 90 to 139 mmHg B. Diastolic Blood Pressure: 60 to 89 mmHg
4. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
5. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serology, urology) and 12-lead ECG results at screening.
6. Those who agree to contraception during the participation of clinical trial
7. Individuals who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.

Exclusion Criteria:

1. Those who received investigational products or participated in bioequivalence tests within 6 months before the first administration of clinical trial drugs.
2. Those who take barbiturate and any related drugs which may cause induction or inhibition of drug metabolism within 1 month before the first administration of investigational products.
3. Those who donated whole blood or apheresis within 2 months or 1 month respectfully, or received blood transfusion within a month.
4. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
5. Those who exceed an alcohol and cigarette consumption than below criteria A. Alcohol: Man- 21 glasses/week, Woman - 14 glasses/week (1 glass: Soju 50mL, Wine 30mL, or beer 250mL) B. Smoking: 20 cigarettes/day
6. Those who have any history of diabetic mellitus, nephropathy, biliary obstruction, shock, angioedema, cardiac insufficiency, dihydropyridine sensitivity, unstable angina, hypothyroidism.
7. Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
8. Those who are deemed insufficient to participate in this clinical study by investigators.
9. Woman who are pregnant or breastfeeding.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-348 | [Time Frame: Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours]
  AUCt: Area under the concentration-time curve from time zero to time
Cmax of CKD-348 | [Time Frame: Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours]
  Cmax: Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
AUCinf of CKD-348 | [Time Frame: Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours]
  AUCinf: Area under the concentration-time curve from zero up to ∞
Tmax of CKD-348 | [Time Frame: Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours]
  Tmax: Time to maximum plasma concentration
T1/2 of CKD-348 | [Time Frame: Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours]
  T1/2: Terminal elimination half-life
AUCt/AUCinf of CKD-348 | [Time Frame: Pre-dose (0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours]
  AUCt/AUCinf

CONTACTS AND LOCATIONS:
Overall Officials: Yook-Hwan Noh, M.D., PhD., Principal Investigator — Study Principal Investigator
Locations (1):
- H Plus Yangji Hospital, Seoul, Gwanak-gu, South Korea